CLINICAL TRIAL: NCT05817903
Title: Phase II Study of Axitinib Intensification Plus Nivolumab Compared to Nivolumab Alone After Induction With Nivolumab Plus Ipilimumab in mRCC Patients Without Previous Complete Response (AxIn Study).
Brief Title: Axitinib Intensification Plus Nivolumab or Nivolumab Alone After Nivolumab Plus Ipilimumab in mRCC Patients
Acronym: AxIn
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Consorzio Oncotech (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AxIn
Record Dates: First submitted 2023-03-14; First posted 2023-04-18 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: mRCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups (ARM A vs ARM B) in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Experimental): Axitinib (starting dose 5 mg BID orally) in addition to nivolumab (lat dose of 480 mg IV every four weeks as per standard clinical practice)
  Interventions: Drug: Axitinib; Drug: Nivolumab
- ARM B (Active Comparator): Nivolumab (flat dose of 480 mg IV every four weeks as per standard clinical practice) after nivolumab plus ipilimumab induction as per standard clinical practice
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Axitinib — Axitinib will be started at the standard dose of 5 mg BID until progression of disease, unacceptable toxicity, patient' or physician' decision.
  Other Names: Inlyta
  Arms: ARM A
Drug: Nivolumab — Nivolumab will be administered at a flat dose of 480 mg IV every four weeks until progression of disease, unacceptable toxicity, patient' or physician' decision

SUMMARY:
This phase II open label trial randomized patients who completed the induction with nivolumab plus ipilimumab without complete response or progressive disease will be randomized 1:1 to receive axitinib in addition to nivolumab (Arm A) or continue with nivolumab alone (Arm B).Treatment will be continued until progression of disease, unacceptable toxicity, patient's refusal, or physician decision whichever occurred first.

DETAILED DESCRIPTION:
The present study aims to demonstrate if the addition of axitinib to nivolumab maintenance after nivolumab plus ipilimumab induction can improve the rate of response considering that the incidence of partial response was 32% and 51% in Checkmate214 and Keynote426 trials respectively.

This study requires 106 patients to show an improvement from 30% to 50% of the incidence of partial responses with a power of 80%, and alpha-error 0.10 (one-side p).

Assuming a drop out of 10%, the final estimated number to enroll should be 118 (59 in arm A and 59 in arm B).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced RCC with predominantly clear-cell subtype and candidate to receive nivolumab after nivolumab plus ipilimumab induction as per standard clinical practice.
2. Completion of the induction of nivolumab and ipilimumab without toxicity ≥ G2 and no complete response or progressive disease.
3. Male or female subjects aged ≥ 18 years
4. Available tumor tissue sample.
5. At least one measurable lesion as defined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
6. Eastern Cooperative Oncology Group performance status 0 or 1.
7. Adequate organ and bone marrow function based upon meeting all of the following laboratory criteria within 10 days before the start of treatment:

   1. Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 GI/L)
   2. Platelets ≥ 100,000/mm3 (≥ 100 GI/L).
   3. Haemoglobin ≥ 9 g/dL (≥ 90 g/L).
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3.0 × upper limit of normal.
   5. Total bilirubin ≤ 1.5 × the upper limit of normal. For subjects with Gilbert's disease ≤ 3 mg/dL (≤ 51.3 µmol/L).
   6. Serum creatinine ≤ 2.0 × upper limit of normal or calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockroft-Gault.
8. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
9. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 5 months after the last dose of study treatment.
10. Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrhoeic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antioestrogens, low body weight, ovarian suppression or other reasons.

Exclusion Criteria:

1. Prior treatment with systemic therapy for advanced RCC with the exclusion of the induction of nivolumab and ipilimumab.
2. Prior adjuvant or neoadjuvant therapy
3. Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis
4. Diagnosis of any non-RCC malignancy occurring within 2 years prior to the date of the start of treatment except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix or low-grade prostate cancer with no plans for treatment intervention.
5. Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before the start of treatment. Systemic treatment with radionuclides within 6 weeks before the start of treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before the start of treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of treatment.
7. Concomitant anticoagulation at therapeutic doses with oral anticoagulants (e.g., warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel).
8. In past 6 months: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack.
9. Chronic treatment with corticosteroids or other immunosuppressive agents (with the exception of inhaled or topical corticosteroids or corticosteroids with a daily dosage equivalent ≤ 10 mg prednisone if given for disorders other than renal cell cancer). Subjects with brain metastases requiring systemic corticosteroid are not eligible.
10. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    I. Cardiovascular disorders:
    1. Symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias.
    2. Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
    3. Stroke (including TIA), myocardial infarction, or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before the start of treatment.

    II. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:
    1. Tumors invading the GI-tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction.
    2. Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before the start of treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed before the start of treatment.

    III. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 3 months before the start of treatment.

    IV. Cavitating pulmonary lesion(s) or known endobronchial disease manifestation.

    V. Lesions invading major pulmonary blood vessels.

    VI. Other clinically significant disorders such as:
    1. Active infection requiring systemic treatment, infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)- related illness, or chronic hepatitis B or C infection.
    2. Serious non-healing wound/ulcer/bone fracture.
    3. Malabsorption syndrome.
    4. Uncompensated/symptomatic hypothyroidism.
    5. Moderate to severe hepatic impairment (Child-Pugh B or C).
    6. Requirement for hemodialysis or peritoneal dialysis.
    7. History of solid organ transplantation.
    8. In past 6 months: deep vein thrombosis or pulmonary embolism.
    9. History of aneurysms and/or artery dissections
11. Major surgery (e.g., GI surgery, removal or biopsy of brain metastasis) within 3 months before the start of treatment. Complete wound healing from major surgery must have occurred 1 month before the start of treatment and from minor surgery (e.g., simple excision, tooth extraction) at least 10 days before the start of treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
12. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 msec within 1 month before the start of treatment (see Section 5.5.4 for Fridericia formula). Three ECGs must be performed. If the average of these three consecutive results for QTcF is ≤ 500 msec, the subject meets eligibility in this regard.
13. Vaccination within 4 weeks of the first dose of nivolumab and while on trials is prohibited except for administration of inactivated vaccines.
14. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
15. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
16. Has a history of substance abuse or medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
17. Has illness or medical conditions that are unstable or could jeopardize the safety of the patient and his or her compliance in the study.
18. Pregnant or lactating females.
19. Inability to swallow tablets or capsules.
20. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
21. Rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of axitinib in addition to nivolumab compared to nivolumab alone at the end of the induction with nivolumab plus ipilimumab in mRCC. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
  The response rate will be evaluated as the number of patients with complete or partial response in each arm. Response rate will be evaluated using RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
  The PFS is defined as the time interval from the date of randomization to the date of radiological or clinical progression or death due to any cause. PFS will be reported as the median value and estimated by Kaplan-Meier method, difference between the two arms will be assessed by log-rank test.
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
  The OS is defined as the time interval from the date of randomization to the date of death due to any cause. OS will be reported as the median value and estimated by Kaplan-Meier method, difference between the two arms will be assessed by log-rank test.
Depth of response. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
  The depth of response is defined as the number of patients who achieved different grades of tumor reduction between the two arms. Difference in the depth of response between will be reported as absolute number and percentage and difference between the two groups will be analyzed.
Duration of response (DOR). | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
  The DOR is the length of time that a tumor continues to respond to treatment without the cancer growing or spreading. DOR will be reported as the median value and estimated by Kaplan-Meier method, difference between the two arms will be assessed by log-rank test.
Health status and life status | From date of enrollment until the date of first documented progression or date of death from any cause
  Quality of life will be evaluated by FKSI-19 and EQ-5D-5L questionnaires within 3 days prior the first study treatment, the first day of each cycle (1, 3, 5, etc.) of nivolumab prior to treatment administration, at the end of treatment visit.
incidence of Treatment-Emergent Adverse Events, Serious adverse events and events of clinical interest, as assessed by the Investigators | all the adverse events occurring from the randomization to 100 days after the last dose of drug
  This analysis will include all the adverse events occurring from the randomization to 100 days after the last dose of drug. Incidence of adverse events will be reported as absolute number and percentage and difference between the two groups will be analyzed.

OTHER OUTCOMES:
expression of PD-L1, PBRM1, CD31 on tumor cells ad CD8+ on lymphocytes | 24 months
  Patients enrolled will be evaluated for the expression in an archival paraffin embedded tumour tissue block for the immunohistochemistry expression of PBRM1, PD-L1, CD31 and immune infiltration CD8+. The expression of these proteins will be related to the main outcomes investigated in the study. Tumor samples will be collected and analyzed at the end of the trial. The analysis will be performed by two expert pathologists in GU tumors at Fondazione Policlinico Universitario Agostino Gemelli IRCCS in Rome, Italy.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Iacovelli, Principal Investigator — Fondazione Policlinico "A. Gemelli", Università Cattolica Sacro Cuore
Locations (23):
- Italy (23):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo
  - Azienda Ospedaliera per l'emergenza Cannizzaro, Catania
  - ASST di Cremona, Cremona
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia - IEO, Milan
  - A.O.U. Policlinico di Modena, Modena
  - Policlinico Duilio Casula - Azienda Ospedaliero-Universitaria di Cagliari, Monserrato
  - Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara
  - Istituto Oncologico Veneto, Padua
  - Casa Di Cura La Maddalena S.P.A., Palermo
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Azienda Ospedalieo-Universitaria Pisana, Pisa
  - San Carlo - Azienda Ospedaliera Regionale, Potenza
  - Presidio Ospedaliero S. Maria Delle Grazie, Pozzuoli
  - IRCCS - AUSL di Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Romano di Lombardia
  - IRCCS - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Integrata Verona - Borgo Roma, Verona
  - Ospedale di Belcolle, Viterbo

IPD SHARING:
Plan to Share IPD: No